CLINICAL TRIAL: NCT00030186
Title: An Open-Label Study of CEP-701 in Patients With Refractory, Relapsed, or Poor Risk Acute Myeloid Leukemia Expressing FLT-3 Activating Mutations
Brief Title: Open Study of CEP-701 in Patients With Refractory Acute Myeloid Leukemia With FLT-3 Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0701a/202/ON/US
Record Dates: First submitted 2002-02-07; First posted 2002-02-08 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Leukemia, Myeloid
Keywords: AML; FLT-3 mutation
MeSH Terms: conditions — Leukemia, Myeloid | interventions — lestaurtinib

ARMS (3):
- Cycle 1 (Experimental): 60mg
  Interventions: Drug: CEP-701 60mg
- Cycle 2 (Experimental): 80mg dependent upon response to Cycle 1
  Interventions: Drug: Cep-701 80mg
- Cycle 2b (Experimental): 40mg dependent upon response to Cycle 1
  Interventions: Drug: Cep-701 40mg

INTERVENTIONS:
Drug: CEP-701 60mg — 60mg orally 2 times a day for 28 days
  Arms: Cycle 1
Drug: Cep-701 80mg — 80mg 2 times a day, dependent upon response to cycle 1
  Arms: Cycle 2
Drug: Cep-701 40mg — 40mg 2 times a day, dependent upon response to cycle 1
  Arms: Cycle 2b

SUMMARY:
The purpose of this study is to determine the response rate of patients with refractory, relapsed or poor risk AML expressing FLT-3 activating mutations, when administered CEP-701 at a dosage of 60 mg 2 times a day.

DETAILED DESCRIPTION:
This is an open-label study of CEP-701 in patients with refractory, relapsed, or poor risk AML expressing FLT-3 activating mutations. Patients who meet eligibility criteria will be enrolled at a dosage of 60 mg orally 2 times a day for 28 days (1 cycle). Upon completion of cycle 1, the dosage may be increased to 80mg 2 times a day or decreased to 40 mg 2 times a day, dependent upon response to 60 mg dosage.

ELIGIBILITY:
INCLUSION CRITERIA:

* patient must have confirmed diagnosis of refractory or relapsed AML that expresses a FLT-3 mutation
* patient must have life expectancy of more than 2 months
* patient must be fully recovered from reversible side effects of previous therapy for cancer

EXCLUSION CRITERIA:

* total bilirubin, ALT or AST greater than 2 times upper limit of normal
* patient <65 years of age with estimated creatinine clearance less than 60 mL/min; patient >65 years of age with serum creatinine > 1.5 times the upper limit of normal (ULN)
* received any investigational drug within past 4 weeks
* GI disturbance/malabsorption that may affect absorption of CEP-701
* HIV positive
* received NSAID within prior 14 days
* has active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2002-01; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Blood Samples and/or bone marrow assessments for complete remission (CR), complete tumor clearance (CTC), or hematologic response (HR) from bone marrow | 56 days
  Response rate of patients with refactory, relapsed, or poor risk acute myeloid leukemia (AML) expressing Fms-like tyrosine kinase 3 (FLT-3) activating mutations. CR is defined as presence of less than 5% myeloblasts in bone marrow with normalized peripheral blood cell counts. HR is defined as a 50% or more decrease in the absolute number of peripheral blast count or at least a 50% reduction in bone marrow blasts.

SECONDARY OUTCOMES:
Number of days to response | 56 Days
  Response as defined by CR, CTC, or HR.
Number of days to disease progression | 56 Days
  Response as defined by CR, CTC, or HR.
Levels of FLT-3 phosphorylation inhibition in vivo | 56 Days
  The degree of inhibition of FLT-3 autophosphorylation measured in ex vivo bioassay plasma samples